CLINICAL TRIAL: NCT02683824
Title: Detection of Integrin Alpha-v-Beta 6 in Pancreatic Cancer With [18F]-R01-MG-F2: a First in Human Study
Brief Title: Integrin Alpha-v-Beta and [18F]-R01-MG-F2 PET/CT in Measuring Response in Patients With Pancreatic Cancer and Healthy Volunteers
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IRB-34376; NCI-2015-01887 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 4593; PANC0020 (Other: OnCore); P30CA124435 (NIH)
Record Dates: First submitted 2016-01-21; First posted 2016-02-17 (Estimated); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Healthy Subject; Pancreatic Carcinoma
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Tomography, X-Ray Computed; Tomography; Positron-Emission Tomography; Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- pancreatic cancer patients (Experimental): Patients receive [18F]FP-R01-MG-F2 IV and undergo PET/CT or PET/MRI scan immediately after and at 60 and 120 minutes.
  Interventions: Diagnostic Test: Computed Tomography; Other: Laboratory Biomarker Analysis; Diagnostic Test: PET/MRI scan; Drug: [18F]FP-R01-MG-F2
- healthy patients (Experimental): Patients receive [18F]FP-R01-MG-F2 IV and undergo PET/CT or PET/MRI scan immediately after and at 60 and 120 minutes.
  Interventions: Diagnostic Test: Computed Tomography; Other: Laboratory Biomarker Analysis; Diagnostic Test: PET/MRI scan; Drug: [18F]FP-R01-MG-F2

INTERVENTIONS:
Diagnostic Test: Computed Tomography — Undergo CT scan
  Other Names: CAT; CAT Scan; Computerized Axial Tomography; Computerized Tomography; CT; CT SCAN; tomography
Other: Laboratory Biomarker Analysis — Correlative studies
Diagnostic Test: PET/MRI scan — Undergo PET/MRI scan
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET SCAN; Positron Emission Tomography; Positron Emission Tomography Scan; Positron-Emission Tomography; magnetic resonance imaging
Drug: [18F]FP-R01-MG-F2 — radioactive tracer

SUMMARY:
This pilot clinical trial studies the use of integrin alpha-v-beta [18F]-R01-MG-F2 Positron Emission Tomography/Computed Tomography (PET/CT) and Positron Emission Tomography-Magnetic Resonance Imaging in (PET/MRI) in measuring response in patients with pancreatic cancer and healthy volunteers. Integrins, such as integrin alpha-v-beta-6 (avb6), are a family of membrane receptors that are overexpressed on the cell surface of pancreatic cancers. [18F]-R01-MG-F2 targets avb6, which may improve early detection of and better stratify treatment options for patients with pancreatic cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Evaluate the biodistribution and safety of [18F]FP-R01-MG-F2 in healthy volunteers.

II. Evaluate the feasibility of [18F]FP-R01-MG-F2 PET/CT scanning in patients with pancreatic cancer.

OUTLINE:

Patients receive [18F]FP-R01-MG-F2 intravenously (IV) and undergo PET/CT or PET/MR scan immediately after and at 60 and 120 minutes. Patients will be followed up at 24-48 hours.

ELIGIBILITY:
Inclusion Criteria:

Healthy volunteers:

1. Must be 18 years of age or older.
2. Must have no known medical problems and have had a full medical exam within 6 months of the study. If healthy volunteers have not had a full medical exam within 6 months of the study, one of the nuclear medicine physicians will conduct the medical exam prior to any study procedures.
3. Must understand and voluntarily have signed an Informed Consent after its contents have been fully explained.
4. Women of child bearing potential (as defined as women who are not post menopausal for 12 months or who have had no previous surgical sterilization) and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation and for 30 days after the last dose.

Pancreatic cancer subjects:

1. Participant must be 18 years or older at the time of radiotracer administration
2. Provides written informed consent
3. Suspected or established diagnosis of pancreatic cancer based on any radiographic scan or pathology and who is scheduled for surgery OR Biopsy proven diagnosis of pancreatic cancer who is no longer a surgical candidate

Exclusion Criteria:

Healthy volunteers:

1. Participant is less than 18 year-old
2. Pregnant or breast feeding women.
3. Patients who are not likely to comply with the protocol requirements.

Pancreatic cancer subjects:

1. Participant is pregnant or breast-feeding
2. Participant is not able to comply with the study procedures
3. Participant has serious uncontrolled concurrent medical illness that would limit compliance with study requirements
4. Metallic implants (contraindicated for MRI)
5. History of renal insufficiency (only for MRI contrast administration)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2016-01-12 (Actual); Primary Completion 2021-09-27 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Biodistribution of [18F]FP-R01-MG-F2 (%ID/g) | Up to 3 hours after tracer injection
  From the Region-of-Interest (ROI) image analysis, the biodistribution data will be reported in percent injected dose per gram of tissue (%ID/g). ROI analysis will be performed on normal brain, thyroid, lungs, mediastinum, liver, spleen, intestines, kidneys, urinary bladder and gluteal muscle.
Biodistribution of [18F]FP-R01-MG-F2 (SUV) | Up to 3 hours after tracer injection
  From the Region-of-Interest (ROI) image analysis, the biodistribution data will be reported in Standardized Uptake Values (SUV). ROI analysis will be performed on normal brain, thyroid, lungs, mediastinum, liver, spleen, intestines, kidneys, urinary bladder and gluteal muscle.
Dosimetry of [18F]FP-R01-MG-F2 (rem/mCi) | Up to 3 hours after tracer injection
  Using the biodistribution data (uptake in %ID/g or SUV), the tracer's complete dosimetry across all organs, tissues or cells will be determined using the OLINDA software. These data will be reported in rem/mCi.
Dosimetry of [18F]FP-R01-MG-F2 (mSv/MBq) | Up to 3 hours after tracer injection
  Using the biodistribution data (uptake in %ID/g or SUV), the tracer's complete dosimetry across all organs, tissues or cells will be determined using the OLINDA software. These data will be reported in mSv/MBq.

CONTACTS AND LOCATIONS:
Overall Officials: Andrei Iagaru, Principal Investigator — Stanford Cancer Institute
Locations (1):
- Stanford University, School of Medicine, Palo Alto, California, United States

REFERENCES:
- [Derived] Nakamoto R, Ferri V, Duan H, Hatami N, Goel M, Rosenberg J, Kimura R, Wardak M, Haywood T, Kellow R, Shen B, Park W, Iagaru A, Gambhir SS. Pilot-phase PET/CT study targeting integrin alphavbeta6 in pancreatic cancer patients using the cystine-knot peptide-based 18F-FP-R01-MG-F2. Eur J Nucl Med Mol Imaging. 2022 Dec;50(1):184-193. doi: 10.1007/s00259-021-05595-7. Epub 2021 Nov 3. PMID 34729628